CLINICAL TRIAL: NCT05240443
Title: Effect of Bariatric Surgery on Chronic Renal Disease (BARICADE): A Pilot Randomized Controlled Trial
Brief Title: Bariatric Surgery and Chronic Renal Disease
Acronym: BARICADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Collaborators: American College of Surgeons (Other); McMaster Surgical Associates (Other)
Responsible Party: Principal Investigator, Dennis Hong MD, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14388-GRA
Record Dates: First submitted 2022-01-17; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Bariatric Surgery; Chronic Kidney Diseases; Obesity
Keywords: Bariatric Surgery; Chronic Kidney Disease; Obesity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Single-centre, open-label, parallel-arm feasibility randomized controlled trial with blinded endpoint assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric Surgery + Medical Management for Chronic Kidney Disease (Experimental): The intervention group will include medical management and bariatric surgery, which will consist of Roux-en-Y gastric bypass or sleeve gastrectomy performed according to local practice standards. Medical management for CKD will be directed by nephrologists at St. Joseph's Healthcare Hamilton. Comorbidities such as hypertension, dyslipidemia, and type 2 diabetes will be managed at the discretion of individual nephrologists. Generally, this can include anti-hypertensives (angiotensin-converting enzyme inhibitors or angiotensin receptor blockers) for systolic blood pressure control below a target of <140/90 mmHg (<130/80 in patients with type 2 diabetes), statins in patients with dyslipidemia to target low-density lipoprotein <2mmol/L for the treatment of CKD.
  Interventions: Procedure: Bariatric Surgery + Medical Management of CKD.
- Medical Management for Chronic Kidney Disease (Active Comparator): Medical management for CKD will be directed by nephrologists at St. Joseph's Healthcare Hamilton. Comorbidities such as hypertension, dyslipidemia, and type 2 diabetes will be managed at the discretion of individual nephrologists. Generally, this can include anti-hypertensives (angiotensin-converting enzyme inhibitors or angiotensin receptor blockers) for systolic blood pressure control below a target of <140/90 mmHg (<130/80 in patients with type 2 diabetes), statins in patients with dyslipidemia to target low-density lipoprotein <2mmol/L for the treatment of CKD.
  Interventions: Other: Medical Management for CKD

INTERVENTIONS:
Procedure: Bariatric Surgery + Medical Management of CKD. — The intervention group will include medical management and bariatric surgery, which will consist of Roux-en-Y gastric bypass or sleeve gastrectomy performed according to local practice standards. Medical management for CKD will be directed by nephrologists at St. Joseph's Healthcare Hamilton. Comorbidities such as hypertension, dyslipidemia, and type 2 diabetes will be managed at the discretion of individual nephrologists. Generally, this can include anti-hypertensives (angiotensin-converting enzyme inhibitors or angiotensin receptor blockers) for systolic blood pressure control below a target of <140/90 mmHg (<130/80 in patients with type 2 diabetes), statins in patients with dyslipidemia to target low-density lipoprotein <2mmol/L for the treatment of CKD.
  Arms: Bariatric Surgery + Medical Management for Chronic Kidney Disease
Other: Medical Management for CKD — Medical management for CKD will be directed by nephrologists at St. Joseph's Healthcare Hamilton. Comorbidities such as hypertension, dyslipidemia, and type 2 diabetes will be managed at the discretion of individual nephrologists. Generally, this can include anti-hypertensives (angiotensin-converting enzyme inhibitors or angiotensin receptor blockers) for systolic blood pressure control below a target of <140/90 mmHg (<130/80 in patients with type 2 diabetes), statins in patients with dyslipidemia to target low-density lipoprotein <2mmol/L for the treatment of CKD.
  Arms: Medical Management for Chronic Kidney Disease

SUMMARY:
Obesity can be a major driver for the development of chronic kidney disease (CKD), which is a leading cause of death and significant loss in quality of life. A growing body of evidence has shown bariatric (metabolic) surgery as a novel approach to reduce the progression of CKD and reduce morbidity with sustained weight loss. This pilot trial will inform the design and execution of a large RCT that could determine the efficacy of bariatric surgery in the treatment of patients with CKD in the context of obesity. Ultimately, the results have the potential to influence guidelines that may deem bariatric surgery as a viable treatment option for CKD and reduce the morbidity from this chronic condition and inform clinical practice.

DETAILED DESCRIPTION:
Obesity is a major driver for the development of CKD, which is a leading cause of death and greatly reduces one's quality of life. With a global prevalence of 9.1% (7.2% in Canada), CKD affects an estimated 13.6% of the American population and was associated with over $50 billion in healthcare costs, with an additional $30 billion in costs associated with end-stage renal disease (ESRD). Moreover, with an aging Canadian population, the prevalence of CKD is expected to rise over the coming years with patients progressing to higher disease burdens. This, in part, has led to a substantial increase in renal replacement therapy by means of dialysis or kidney transplant by 43.1% since 1990. Obesity is also an important modulatory factor in the development of poor outcomes as a result of CKD and has been linked to an increased rate of progression from CKD towards kidney failure. The most common comorbidities in patients with CKD were hypertension, diabetes, heart failure, chronic pulmonary disease, and atrial fibrillation and in Canada, 25% of patients with CKD have at least 3 or more comorbidities which too are associated with an increased risk of hospitalization and early death. Most worryingly, unlike other non-communicable diseases today, the age-standardized mortality for CKD has not declined over the past decades. Therefore, innovative strategies are of timely importance to reduce mortality and morbidity in patients with CKD and thus urgently needed, especially in patients with multiple comorbidities and targeting weight loss is a promising avenue to find novel treatment options.

Bariatric surgery has been shown to not only facilitate sustained weight loss in patients with obesity, but also independently improve cardiac risk factors such as dyslipidemia, hypertension, and type 2 diabetes mellitus. It has also been shown to reverse glomerular hyperfiltration and lower proteinuria in patients with obesity and normal kidney function and delay the need for renal transplantation in patients with ESRD. Moreover, the protective benefit of bariatric surgery has been shown to reduce risk of CKD progression for up to seven years after intervention in observational studies. However, current guidelines do not address a role for bariatric surgery in the management of patients with obesity and CKD.

Given the poor outcomes with patients with obesity and CKD, a RCT to assess the efficacy and safety of bariatric surgery as an intervention for patients with CKD is of timely importance. The present proposed pilot RCT of bariatric surgery versus medical management alone for patients with morbid obesity and CKD in order to assess whether a large, multi-centre, efficacy trial is feasible. The results of the proposed pilot study will thus inform the design of a larger RCT in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patient age >18
* Body mass index > 40 (or > 35 kg/m2 for patients with comorbidities)
* Diagnosis of CKD stage III (G3a or A2) defined as the presence of any of the following:

  1. glomerular filtration rate (GFR) under 60 mL/min/1.73 m2 as estimated from serum creatinine or cystatin C with the CKD-EPI equation
  2. ACR > 30 mg/g
* Patient is deemed eligible to undergo bariatric surgery according to Ontario Bariatric Network (OBN) guidelines [contradictions to OBN guidelines include non-Ontario resident, age >70 years, history of cancer <2 years, current substance use disorder, accessed palliative care, previous organ transplant (liver, heart, or lungs), active cardiac disease, major revascularization procedures within 6 months, or severe liver disease with ascites <1 year]

Exclusion Criteria:

* Hospital admission for kidney failure or acute kidney injury within 30 days of enrollment
* Documented GFR > 60 mL/min/1.73 m2 or ACR < 30 mg/g within 30 days of enrollment
* Documented confounders of kidney function measurement such as urinary tract infection or use of creatinine elevating medications or use of medications which interfere with measurement
* Contradiction to OBN guidelines including non-Ontario resident, age >70 years, history of cancer <2 years, current substance use disorder, accessed palliative care, previous organ transplant (liver, heart, or lungs), active cardiac disease, major revascularization procedures within 6 months, or severe liver disease with ascites <1 year
* Life expectancy <2 years due to non-CKD causes OR Untreated or inadequately treated psychiatric illness OR Risk of general anesthesia deemed too excessive OR Inability to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Estimated Glomerular Filtration Rate (units: ml/min/1.73m2) at 6 months | Month 6
Estimated Glomerular Filtration Rate (units: ml/min/1.73m2) at 12 months | Month 12
Estimated Glomerular Filtration Rate (units: ml/min/1.73m2) at 18 months | Month 18
Measured Glomerular Filtration Rate (units: ml/min/1.73m2) at 6 months | Month 6
Measured Glomerular Filtration Rate (units: ml/min/1.73m2) at 12 months | Month 12
Measured Glomerular Filtration Rate (units: ml/min/1.73m2) at 18 months | Month 18
Creatine Clearance (units: mL/min) at 6 months | Month 6
Creatine Clearance (units: mL/min) at 12 months | Month 12
Creatine Clearance (units: mL/min) at 18 months | Month 18
Serum Creatinine (units: μmol/L) at 6 months | Month 6
Serum Creatinine (units: μmol/L) at 12 months | Month 12
Serum Creatinine (units: μmol/L) at 18 months | Month 18
Serum Cystatin C (units: mg/L) at 6 months | Month 6
Serum Cystatin C (units: mg/L) at 12 months | Month 12
Serum Cystatin C (units: mg/L) at 18 months | Month 18
Urine Albumin-Creatine Ratio (units: mg/g) at 6 months | Month 6
Urine Albumin-Creatine Ratio (units: mg/g) at 12 months | Month 12
Urine Albumin-Creatine Ratio (units: mg/g) at 18 months | Month 18

SECONDARY OUTCOMES:
Weight and height will be combined to report BMI in kg/m^2 at 6 months | Month 6
Weight and height will be combined to report BMI in kg/m^2 at 12 months | Month 12
Weight and height will be combined to report BMI in kg/m^2 at 18 months | Month 18
Recruitment Rate (60 patients will be recruited at an average recruitment rate of 1.25 patients per site per month.) | Month 6
  60 patients will be recruited at an average recruitment rate of 1.25 patients per site per month.
Intervention Administration Rate | Month 6
  >80% of patients randomized to the intervention arm will undergo bariatric surgery within 30 days of randomization.
Crossover rate between control and intervention arm | Month 6
Number of patients adhering to study treatments | Month 6
  Patients will be monitored and asked about adherence at follow-ups.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hong, MD MSc FRCSC, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saran R, Robinson B, Abbott KC, Agodoa LY, Albertus P, Ayanian J, Balkrishnan R, Bragg-Gresham J, Cao J, Chen JL, Cope E, Dharmarajan S, Dietrich X, Eckard A, Eggers PW, Gaber C, Gillen D, Gipson D, Gu H, Hailpern SM, Hall YN, Han Y, He K, Hebert H, Helmuth M, Herman W, Heung M, Hutton D, Jacobsen SJ, Ji N, Jin Y, Kalantar-Zadeh K, Kapke A, Katz R, Kovesdy CP, Kurtz V, Lavalee D, Li Y, Lu Y, McCullough K, Molnar MZ, Montez-Rath M, Morgenstern H, Mu Q, Mukhopadhyay P, Nallamothu B, Nguyen DV, Norris KC, O'Hare AM, Obi Y, Pearson J, Pisoni R, Plattner B, Port FK, Potukuchi P, Rao P, Ratkowiak K, Ravel V, Ray D, Rhee CM, Schaubel DE, Selewski DT, Shaw S, Shi J, Shieu M, Sim JJ, Song P, Soohoo M, Steffick D, Streja E, Tamura MK, Tentori F, Tilea A, Tong L, Turf M, Wang D, Wang M, Woodside K, Wyncott A, Xin X, Zang W, Zepel L, Zhang S, Zho H, Hirth RA, Shahinian V. US Renal Data System 2016 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2017 Mar;69(3 Suppl 1):A7-A8. doi: 10.1053/j.ajkd.2016.12.004. No abstract available. PMID 28236831
- [Background] Coresh J, Selvin E, Stevens LA, Manzi J, Kusek JW, Eggers P, Van Lente F, Levey AS. Prevalence of chronic kidney disease in the United States. JAMA. 2007 Nov 7;298(17):2038-47. doi: 10.1001/jama.298.17.2038. PMID 17986697
- [Background] Bello AK, Ronksley PE, Tangri N, Kurzawa J, Osman MA, Singer A, Grill A, Nitsch D, Queenan JA, Wick J, Lindeman C, Soos B, Tuot DS, Shojai S, Brimble S, Mangin D, Drummond N. Prevalence and Demographics of CKD in Canadian Primary Care Practices: A Cross-sectional Study. Kidney Int Rep. 2019 Jan 21;4(4):561-570. doi: 10.1016/j.ekir.2019.01.005. eCollection 2019 Apr. PMID 30993231
- [Background] GBD Chronic Kidney Disease Collaboration. Global, regional, and national burden of chronic kidney disease, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2020 Feb 29;395(10225):709-733. doi: 10.1016/S0140-6736(20)30045-3. Epub 2020 Feb 13. PMID 32061315
- [Background] Eknoyan G. Obesity and chronic kidney disease. Nefrologia. 2011;31(4):397-403. doi: 10.3265/Nefrologia.pre2011.May.10963. Epub 2011 May 30. PMID 21623393
- [Background] Tonelli M, Wiebe N, Guthrie B, James MT, Quan H, Fortin M, Klarenbach SW, Sargious P, Straus S, Lewanczuk R, Ronksley PE, Manns BJ, Hemmelgarn BR. Comorbidity as a driver of adverse outcomes in people with chronic kidney disease. Kidney Int. 2015 Oct;88(4):859-66. doi: 10.1038/ki.2015.228. Epub 2015 Jul 29. PMID 26221754
- [Background] Cockwell P, Fisher LA. The global burden of chronic kidney disease. Lancet. 2020 Feb 29;395(10225):662-664. doi: 10.1016/S0140-6736(19)32977-0. Epub 2020 Feb 13. No abstract available. PMID 32061314
- [Background] Docherty NG, le Roux CW. Bariatric surgery for the treatment of chronic kidney disease in obesity and type 2 diabetes mellitus. Nat Rev Nephrol. 2020 Dec;16(12):709-720. doi: 10.1038/s41581-020-0323-4. Epub 2020 Aug 10. PMID 32778788
- [Background] Schauer PR, Kashyap SR, Wolski K, Brethauer SA, Kirwan JP, Pothier CE, Thomas S, Abood B, Nissen SE, Bhatt DL. Bariatric surgery versus intensive medical therapy in obese patients with diabetes. N Engl J Med. 2012 Apr 26;366(17):1567-76. doi: 10.1056/NEJMoa1200225. Epub 2012 Mar 26. PMID 22449319
- [Background] Chagnac A, Weinstein T, Herman M, Hirsh J, Gafter U, Ori Y. The effects of weight loss on renal function in patients with severe obesity. J Am Soc Nephrol. 2003 Jun;14(6):1480-6. doi: 10.1097/01.asn.0000068462.38661.89. PMID 12761248
- [Background] Al-Bahri S, Fakhry TK, Gonzalvo JP, Murr MM. Bariatric Surgery as a Bridge to Renal Transplantation in Patients with End-Stage Renal Disease. Obes Surg. 2017 Nov;27(11):2951-2955. doi: 10.1007/s11695-017-2722-6. PMID 28500419
- [Background] Friedman AN, Wahed AS, Wang J, Courcoulas AP, Dakin G, Hinojosa MW, Kimmel PL, Mitchell JE, Pomp A, Pories WJ, Purnell JQ, le Roux C, Spaniolas K, Steffen KJ, Thirlby R, Wolfe B. Effect of Bariatric Surgery on CKD Risk. J Am Soc Nephrol. 2018 Apr;29(4):1289-1300. doi: 10.1681/ASN.2017060707. Epub 2018 Jan 15. PMID 29335242
- [Background] Friedman AN, Miskulin DC, Rosenberg IH, Levey AS. Demographics and trends in overweight and obesity in patients at time of kidney transplantation. Am J Kidney Dis. 2003 Feb;41(2):480-7. doi: 10.1053/ajkd.2003.50059. PMID 12552513
- [Background] Bolignano D, Zoccali C. Effects of weight loss on renal function in obese CKD patients: a systematic review. Nephrol Dial Transplant. 2013 Nov;28 Suppl 4:iv82-98. doi: 10.1093/ndt/gft302. Epub 2013 Oct 2. PMID 24092846